CLINICAL TRIAL: NCT05822518
Title: Outcome of Perioperative Immune Enhancing Nutrition in Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Ammar Fathi Mohamed AlOrabi, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nutrition in R.cystectomy
Record Dates: First submitted 2023-04-01; First posted 2023-04-20 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Cancer, Bladder; Cystostomy; Complications
Keywords: radical cystectomy; complications; immune-nutrition; immune enhancing nutrition; bladder cancer; muscle invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional protocol group (No Intervention): patients who are enrolled in conventional pre and post operative routine preparation for surgery protocol.
- immune enhancing nutrition protocol group (Active Comparator): patients who are enrolled in pre and post operative routine preparation for surgery protocol plus immune enhancing nutrition administration pre and post operatively.
  Interventions: Dietary Supplement: Neo-mune powder (otsuka pharmaceutical); Drug: Dipeptiven solution (Fresenius Kabi pharmaceutical)

INTERVENTIONS:
Dietary Supplement: Neo-mune powder (otsuka pharmaceutical) — * Preoperative: Neo-mune (otsuka pharmaceutical) powder 60 gm o.d. orally (contains glutamine, arginine and fish oil) for 3 days.
  * Postoperative: Neo-mune (otsuka pharmaceutical) powder 60 gm o.d. orally (contains glutamine, arginine and fish oil) for 2 weeks starting when the intestinal sounds are audible.
  Arms: immune enhancing nutrition protocol group
Drug: Dipeptiven solution (Fresenius Kabi pharmaceutical) — Dipeptiven (Fresenius Kabi pharmaceutical) solution 50 mg o.d IV ( contains L-ananyl-L-glutamine dipeptide) post operatively for 5 days starting from the operation day.
  Arms: immune enhancing nutrition protocol group

SUMMARY:
The aim of this study is to evaluate the outcome of perioperative immune-nutrition with glutamine, arginine and fish oil in patients undergoing radical cystectomy as regards to enhancement of healing, increasing immunity and improving overall health status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CT showing bladder mass with radiological staging of T2 or T3.
2. Patients pathologically proven to have cancer bladder.
3. Patients undergoing radical cystectomy with ileal conduit.
4. The American Society of Anesthesiologists Physical Status classification system (ASA PS) of 1, 2 or 3.

Exclusion Criteria:

1. Coagulopathy.
2. Distant metastasis.
3. Body mass index less than 18.5.
4. Relevant food allergies.
5. Severe renal and hepatic insufficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  The number of postoperative complications, either infectious or non-infectious. Postoperative complications will be assessed and classified according to modified Clavien-Dindo classification. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V) in which grade I represents the least severe complications and grade V represents the most severe complications.
Wound healing | 30 days
  The number of properly healed wounds. wound healing will be assessed by Pressure Ulcer Scale for Healing (PUSH) tool. this tool give every wound a score depending on surface area, exudate amount and tissue type. the scoring system ranging from 0 to 17 in which "0" represents completely healed wound and "17" represents the least healed wound. Surgical wounds are acute wounds that closure expected timeframe is about 4 weeks.
infectious complications | 30 days
  infection rate will be assessed by need for intervention or prescription of non-prophylactic antibiotics or presence of systemic inflammatory response syndrome (SIRS).

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  will be measured by number of days of hospital stay.
Length of ICU stay | 30 days
  will be measured by number of days of ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt